CLINICAL TRIAL: NCT03755180
Title: The Effectiveness of Exercise Training in Venous Insufficiency
Brief Title: Exercise Training in Venous Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Saliha Gürdal Karakelle, Research Assisstant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 99984023-302.14.04-
Record Dates: First submitted 2018-11-23; First posted 2018-11-27 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Venous Insufficiency
Keywords: Venous Insufficiency; Exercise; Compression Bandages; Duplex Doppler Ultrasonography
MeSH Terms: conditions — Venous Insufficiency; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Exercise Group
  Interventions: Other: Exercise Training; Other: Compression Therapy
- Group 2 (Active Comparator): Compression Group
  Interventions: Other: Compression Therapy

INTERVENTIONS:
Other: Exercise Training — In exercise training, aerobic exercise and strengthening exercises, especially for gastrocnemius and tibialis anterior muscles, will be applied to the patients. In addition the exercise training, Compression Therapy is applied to patients.
  Arms: Group 1
Other: Compression Therapy — Compression therapy is a treatment applied to patients in the form of Four Layer Compression Bandage and Compression Stocking. Four Layer Compression Bandage is a treatment that requires four different types of bandages. The compression stocking is an elastic stock with various tension and length.

SUMMARY:
The aim of this study is to evaluate the effects of exercise training in addition to compression therapy on clinical severity, vein diameter, reflux and quality of life in venous insufficiency patients.

DETAILED DESCRIPTION:
Volunteers who have been diagnosed with venous insufficiency according to the criteria of inclusion, who applied to Istanbul University Istanbul Medical Faculty Cardiovascular Surgery Department will be included this study.

Participants will be randomly allocated 2 groups using the 'Research Randomizer' website. In both groups, a common evaluation protocol will be applied to the patients.

Exercise training in addition to compression bandages will be applied to first group, compression bandages will be applied to second group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of venous insufficiency with duplex ultrasonography
* Classification of CEAP (Clinical-Etiological-Anatomical-Pathological) used in venous insufficiency is C3-C4-C5-C6
* Ankle-brachial index (ABI) is less than 0.7
* Possibility to communicate in written and verbal in Turkish
* Have a level of cognitive ability to understand the instructions given

Exclusion Criteria:

* Presence of deep vein thrombosis
* Ulceration or open burn wound in lower extremity greater than 4 cm
* Presence of infected ulceration
* Cardiorespiratory insufficiency
* Orthopedic, rheumatologic or neurological comorbidities restrain the exercise in lower extremity
* Presence of a psychiatric illness requiring the use of prescribed medicines

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
Chronic Venous Disease Quality of Life Questionnaire (CIVIQ) 20 | Change from Baseline Quality of Life at 6 weeks.
  CIVIQ 20 is a disease-related quality of life assessment form especially for chronic venous insufficiency patients. The total score is at least 0 and at most 100, and the higher scores indicate better quality of life.

SECONDARY OUTCOMES:
Duplex Ultrasonography | Duplex Ultrasonography results is evaluated at baseline and six weeks rehabilitation program.
  Duplex Ultrasonography is a form of ultrasound that produces images that differentiate between the body's soft tissues and its fluid-filled structures. Duplex Ultrasonography provides information on vascular diameter and reflux in chronic venous insufficiency patients.
Venous Clinical Severity Score (VCSS) | Assessment is performed at baseline and six weeks rehabilitation program.
  The VCSS was subsequently developed as an evaluative instrument that would be responsive to changes in disease severity over time and in response to treatment.The total score is at least 0 and at most 30, and the low scores are positively correlated with the severe clinical condition.
Visual Analogue Scale (VAS) | Assessment is performed at baseline and six weeks rehabilitation program.
  The levels of pain felt rest/activity/night will be measured using visual analogue scale (VAS). Patients will be asked to evaluate their pain status with a 10-point scale and high scores are positively correlated with pain.
The 6 Minute Walk Test | Assessment is performed at baseline and six weeks rehabilitation program.
  The 6-min walk test (6 MWT) is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes.
10-Meter Walk Test | Assessment is performed at baseline and six weeks rehabilitation program.
  The 10mWT is used to assess walking speed in meters/second (m/s) over a short distance.
Assessment of Muscle Strength with Handheld Dynamometer | Assessment is performed at baseline and six weeks rehabilitation program.
  The muscle strength of the gastrocnemius and tibialis anterior muscles will be evaluated using the handheld dynamometer.
Short Form 36 (SF-36) | Assessment is performed before treatment and after six weeks rehabilitation program.
  SF-36 is used to assess physical and mental health-related quality of life. The total score is at least 0 and at most 100, and the high scores are positively correlated with the high quality of life.
Measurement of Calf Girth | Assessment is performed at baseline and six weeks rehabilitation program.
  Circumference measurements will be recorded at 10 cm intervals of both lower legs.

CONTACTS AND LOCATIONS:
Overall Officials: Saliha Gürdal, Principal Investigator — Istanbul University Health Sciences Institute; İpek Yeldan, Study Director — Istanbul University Faculty of Health Science
Locations (1):
- Istanbul Faculty of Medicine, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No